CLINICAL TRIAL: NCT05371327
Title: Use of Public Deliberation in Diverse Communities to Improve Consent Processes for Clinical Research
Brief Title: Community Solutions to Adolescent Research Consent - Minor Consent for Biomedical HIV Research
Acronym: C-START
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Amelia Knopf, Associate Professor, Indiana University
Other Study IDs: ME-2018C3-14766
Record Dates: First submitted 2022-03-29; First posted 2022-05-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Informed Consent; HIV Infections
Keywords: Public Deliberation
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Public Deliberants: Minors and adults recruited through a community outreach process.
  Interventions: Behavioral: Public deliberation

INTERVENTIONS:
Behavioral: Public deliberation — Public deliberation is a method for engaging the public in collective decision-making. Its goal is to facilitate debate and discussion that: 1) fosters the formation of reasonable and informed opinions, 2) permits participants to revise their perspectives and positions in light of new information and dialogue with others, and 3) encourages participants to consider not only their own preferences but also the greater goal of a policy or resolution that is justifiable for all persons affected by the issue under debate.

SUMMARY:
Public deliberation is a novel method for engaging the public in collective decision-making. Its goal is to facilitate debate and discussion that: 1) fosters the formation of reasonable and informed opinions, 2) permits participants to revise their perspectives and positions in light of new information and dialogue with others, and 3) encourages participants to consider not only their own preferences but also the greater goal of a policy or resolution that is justifiable for all persons affected by the issue under debate. Public deliberation involves: in-depth education on the topic of interest, presentation of conflicting perspectives from expert witnesses and key stakeholders, facilitated public discussion of core issues, and development of resolutions that are acceptable to participants. Public deliberation requires significant commitment from deliberants who are actively engaged over the course of several sessions. Public deliberation can be successful when more traditional methods of stakeholder engagement fail, as it allows for in-depth discussion and demonstrated awareness of the moral difference in deciding for oneself and others.

Minor consent to biomedical HIV prevention research highlights difficulties with consent, particularly for minors, and how key ethical principles may come into conflict. Typically, institutions and investigators rely upon parental permission to protect minors from research-related harm and coercion. However, the parent permission model may be harmful in stigmatizing health research such as HIV. The consent process creates potential for disclosure of the minor's sensitive behaviors and/or identities to their parents who were otherwise unaware of them. This risk is heightened for sexual and gender minority adolescents, who may face physical and social harm when their sexual or gender identities are disclosed. This risk of harm, and the ethical conflict it creates has contributed to delays in clinical trials and clinical use of HIV prevention methods in minors.

This project will test public deliberation as a method for improving consent processes for engaging individuals from marginalized communities in clinical research on sensitive or stigmatizing health problems. The investigators use minor consent for biomedical HIV prevention research as an exemplar case. The primary hypothesis is that public deliberation will produce a resolution to ethical conflicts in minor consent that is better or different from the results of more traditional study approaches (e.g. surveys, in depth interviews).

ELIGIBILITY:
Inclusion Criteria - Deliberants must:

* Complete the screening survey;
* Be at least 14 years of age;
* Speak and understand English; and,
* Be able to commit to attend all virtual deliberation sessions in their entirety.
* Be one of the following:

  * 14-21years old
  * Have an adolescent who lives with you
  * Closely involved with an adolescent on a regular basis (e.g. grandparent, adult sibling)
  * Work for an organization or program that is invested in the wellbeing of adolescents in your community (e.g. social worker, high school teacher, nonprofit work)
  * Part of an organization or program that is invested in the wellbeing of adolescents in your community (e.g. mentor, volunteer, church youth group)

Exclusion Criteria:

* Those who are obviously inebriated or high at the time of screening, the deliberation event, or the pre-/post-event interviews;
* Those who reside in a home with another eligible participant

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Deliberants will include both adolescents/young adults and adults. They need to live, work, or engage with communities with youth at risk for HIV. Communities can be geographic communities, LGBTQ communities, Black or Latinx communities, etc.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Acceptability of parental permission in consent for HIV biomedical prevention research. | Duration of public deliberation (2-4 weeks)
  One of three items adapted from a previous study (see citation), and are scored separately on a 1-5 scale with 5 being the most acceptable:
  Imagine a teen wants to join a biomedical HIV prevention study like the one you just read about. The teen asks their parent/guardian to come to the research clinic with them. The parent/guardian is given information about the study, and has the opportunity to ask any questions they want to ask. After the parent's questions are answered, they are asked whether or not they give permission for their teen to join the study.
  In this approach to consent, the parent/guardian has the final say about whether the teen can join the study. How acceptable is this approach to research consent?
  1. Completely unacceptable
  2. Somewhat unacceptable
  3. Neither unacceptable nor acceptable
  4. Somewhat acceptable
  5. Completely acceptable
Acceptability of minor self-consent for HIV biomedical prevention research. | Duration of public deliberation (2-4 weeks)
  One of three items adapted from a previous study (see citation), and scored separately on a 1-5 scale with 5 being the most acceptable:
  Imagine again that a teen wants to join a biomedical HIV prevention study like the one you just read about. The teen comes to the research clinic on their own. They read the consent form, and have an opportunity to ask questions. Once their questions are answered, the teen is ready to consent to the study. They are allowed to sign the consent form and join the study without speaking to anyone else about the decision.
  In this approach to consent, the teen is allowed to make the decision about joining the research study on their own. How acceptable is this approach to research consent?
  1. Completely unacceptable
  2. Somewhat unacceptable
  3. Neither unacceptable nor acceptable
  4. Somewhat acceptable
  5. Completely acceptable
Acceptability of ombudsman for consent for HIV biomedical prevention research. | Duration of public deliberation (2-4 weeks)
  Third item, scored 1-5, with 5 most acceptable. Imagine a teen wants to join a biomedical HIV prevention study like the one you just read about. The teen comes to the research clinic on their own. They read the consent form, and have an opportunity to ask questions. The teen is required to have an adult's permission to sign up for the study. They can choose to ask either their parent or a neutral adult, called an "ombudsman." The ombudsman is not in charge of the study; the ombudsman's job is to ensure the teen understands the research study, and to help them think about the risks and benefits of joining the study. The teen would need either their parents' permission OR the ombudsman's permission to join the study.
  In this approach to consent, the teen must have an adult's permission to join the study; the teen would be able to choose whether to seek permission from their parent or the ombudsman. How acceptable is this approach to research consent? (Same 5 responses as above)

SECONDARY OUTCOMES:
Quality of public deliberation | Duration of public deliberation (2-4 weeks)
  This qualitative assessment of transcripts of the public deliberation assesses 4 dimensions of quality (adapted from DeVries, PMID 20378225). This is a group-level measure (rather than individual level). (1) Equal participation is a count of the number and length of comments from participants in transcripts. (2) Respect for opinions of others is a qualitative assessment that includes recognition of value of comments or support. We will assess number of instances and examples. (3) Adoption of a societal perspective is a qualitative assessment of whether opinions or recommendations are from an individual perspective or societal perspective. (4) Reasoned justification of ideas is a qualitative assessment of whether reasons are given when opinions or statements. We will create a scoring rubric for these 4 dimensions specific to the topic of the deliberation, with examples. This is a qualitative description of how the dimension has been met, rather than a numeric score.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Knopf, PhD RN MPH, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine and School of Nursing, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified full data package will be available from principal investigators, including protocol, participant-level quantitative data, public deliberation transcripts, analysis plan, documentation of IRB approval and supporting information listed below.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: up to 7 years after conclusion of study and acceptance of final report by PCORI
Access Criteria: Contact principal investigators, Mary A. Ott MD MA (maott@iu.edu) and Amy S. Knopf PhD MPH RN (asknopf@iu.edu).

REFERENCES:
- [Background] Knopf A, Ott MA, Draucker CB, Fortenberry JD, Reirden DH, Arrington-Sanders R, Schneider J, Straub D, Baker R, Bakoyannis G, Zimet GD. Innovative Approaches to Obtain Minors' Consent for Biomedical HIV Prevention Trials: Multi-Site Quasi-Experimental Study of Adolescent and Parent Perspectives. JMIR Res Protoc. 2020 Mar 30;9(3):e16509. doi: 10.2196/16509. PMID 32224493
- [Background] De Vries R, Stanczyk A, Wall IF, Uhlmann R, Damschroder LJ, Kim SY. Assessing the quality of democratic deliberation: a case study of public deliberation on the ethics of surrogate consent for research. Soc Sci Med. 2010 Jun;70(12):1896-1903. doi: 10.1016/j.socscimed.2010.02.031. Epub 2010 Mar 16. PMID 20378225